CLINICAL TRIAL: NCT01545921
Title: Evaluation and Validation of Quality Of Life Scales in Palliative Advanced Cancer
Brief Title: Cancer End Of Life Evaluation
Acronym: CEOLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of inclusions without reaching the expected number of patients
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CPP-435; 2010-A00196-33 (Other: French Health Products Safety Agency)
Record Dates: First submitted 2011-03-16; First posted 2012-03-07 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2020-11

CONDITIONS: Advanced Cancer
Keywords: Quality Of Life; Cancer; End of life; palliative setting
MeSH Terms: conditions — Neoplasms; Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (Experimental): Patients will complete QoL questionnaires in the following order :
  MVQOLI, then QLQ-C15-PAL, then QUAL-E, evaluation every month until death
  Interventions: Other: Quality Of Life questionnaires completion
- Arm B (Experimental): Patients will complete QoL questionnaires in the following order :
  QLQ-C15-PAL, then MVQOLI, then QUAL-E, evaluation every month until death
  Interventions: Other: Quality Of Life questionnaires completion
- Arm C (Experimental): Patients will complete QoL questionnaires in the following order :
  MVQOLI, then QLQ-C15-PAL, then QUAL-E, evaluation every month and spontaneous QoL completion, until death
  Interventions: Other: Quality Of Life questionnaires completion
- Arm D (Experimental): Patients will complete QoL questionnaires in the following order :
  QLQ-C15-PAL, then MVQOLI, then QUAL-E, evaluation every month and spontaneous QoL completion, until death.
  Interventions: Other: Quality Of Life questionnaires completion

INTERVENTIONS:
Other: Quality Of Life questionnaires completion — Before randomization, all patients will have to complete questionnaires in this order : QLQ-C15-PAL, MVQOLI and QUAL-E.
  MVQOLI and QUAL-E will be completed again 3 days after the first completion at baseline. After this second QoL assessment, the order will be modified according to patient's randomisation : arm A, B, C or D.

SUMMARY:
The aim of this study is to culturally adapt and to validate Quality Of Life tools dedicated to the end of life for French cancer patients.

DETAILED DESCRIPTION:
French clinical research in palliative care is confronted with a lack of tools allowing to estimate in a standardized way a patient related outcome. Scales used today are not specifically adapted to quality of life (QoL) at the end of life patient evaluation. So all the relative dimensions to this disease stage are not estimated. What establishes a brake in the improvement of a quality support.

The dimensions of pain, psychological distress, fatigue, decrease of the autonomy are essential points estimated in "classic" questionnaires and frequently used at the palliative disease stage. However the end of life also recovers the domains of the spirituality, oneself's completion, relationship. These elements are essential to dread better QoL at end of life, but are not or do not little approach on the French questionnaires.

The Missoula-Vitas Quality Of Life Index is a questionnaire developed by Byock, Merriman and Kinzbrunner and specifically designed for palliative situations [I. Byock, 1998]. This QoL tool provides an exhaustive assessment of important dimensions in this setting. The short version is composed of 15 items and asks patients to evaluate 5 dimensions: symptoms, function, interpersonal relationships, well-being and transcendence [I. Byock, 1998].

Another tool, the QUAL-E, is longer with 25 items concerning 5 domains: life completion, relations with the health care system, preparation for end of life, symptom severity and affective social support [KE. Steinhauser, 2002]. However, these QoL tools have not been translated and adapted to French. Another concern is that the lack of specificity for cancer patients.

The first step to improve evaluation of how French patients feel about this phase of their disease is to translate these specific end of life QoL tools. Assessing QoL at the end of life with dedicated tools could help to compare therapeutic strategies and could result in improvements in palliative care.

ELIGIBILITY:
Inclusion Criteria:

* Palliative advanced cancer patient (Palliative chemotherapy, analgesic radiotherapy, surgery of comfort accepted).
* All cancer locations and cancer type
* Patient having the knowledge of their palliative disease stage.
* Patient follow-up at least once a month by a palliative caregiver.
* Age > or = 18 years.
* Dated and signed consent.
* PS > or = 2
* Life expectation > or = 1 month.

Exclusion Criteria:

* Psychiatric Disease or cognitive disorders disrupting the trial understanding and the enlightened and voluntary consent character.
* Patient who can not submit itself to the formal follow-up for psychological, social, family or geographical reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2011-11-11 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Psychometric validation of QUALE and Missoula Vitas Quality Of Life Index (MVQOLI) | Up to 3 years
  Both QUALE and MVQOLI have many questions, and each question is evaluated by a number of points. At the end of completion, a score is calculated thanks to number of points and is used to compare the different times completion :
  * no change of score between the 2 first completion (reproductibility)
  * change score with baseline
  * correlation with QLQ-C15 PAL Score
  * correlation with clinical measure (PS, PPS)

SECONDARY OUTCOMES:
Change in Quality of Life at different times | Up to 3 years
  Every month or more, QUALE, MVQOLI and QLQ-C15-PAL will be completed by patient, a final score will be calculated and compared at different times.
Number of spontaneous questionnaire completions | Up to 3 years
  In arms C and D, patients can complete QLQ-C15-PAL and MVQOLI questionnaires at home if they need it. The number of spontaneous questionnaires completions will be evaluated and the impact on quality of life assessed thanks to calculated score.
Rate of completion | Up to 3 years
  Every month or more, the 3 questionnaires QUALE, MVQOLI and QLQ-C15-PAL have to be completed by patient. The rate of completion will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Commer, MD, Principal Investigator — Institut Cancerologie de l'Ouest
Locations (10):
- France (10):
  - CHU, Angers
  - ICO Paul Papin, Angers
  - CHU Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Hospitalier, Cholet
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Val d'Aurelle Paul Lamarque, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Poirier AL, Kwiatkowski F, Commer JM, D'Aillieres B, Berger V, Mercier M, Bonnetain F. Health-related quality of life in cancer patients at the end of life, translation, validation, and longitudinal analysis of specific tools: study protocol for a randomized controlled trial. Trials. 2012 Apr 20;13:39. doi: 10.1186/1745-6215-13-39. PMID 22520742